CLINICAL TRIAL: NCT05299294
Title: Observational Study of the Use of 8% Capsaicin Patch in Children 0 to 18 Years
Brief Title: Observational Study of the Use of 8% Capsaicin Patch in Children 0 to 18 Years Old
Acronym: CAPSULE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Fondation de France (Other); Fondation Apicil (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0184 (CAPSULE)
Record Dates: First submitted 2021-12-23; First posted 2022-03-29 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Neuropathic Pain; Chronic Pain
Keywords: Neuropathic Pain; Pediatric; Capsaicin
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Data collection — Collecting data on children receiving capsaicine 8% patch for localized neuropathic pain

SUMMARY:
Patients aged less than 18-y with validated 8% capsaicin patch treatment in routine healthcare will be offered to participate the study. If they accept it as well as their parents, they will be included in the study .

Medical data will be recorded and at home, the child or his family will collect pain assessment data.

Tolerance will be monitored at home by phone call from investigational team every 24 hours until normalization. (Less than 24 hours for 75%, 100% to 72 hours on unpublished personal series.) Children will be assessed via scales at inclusion and 1-month, 3-month and 6-month.

DETAILED DESCRIPTION:
Children and teenagers aged less than 18-y, with chronic localized neuropathic pain, may be treated by capsaicin 8% patch. If this indication is validated in pediatric chronic pain consultation, they will be offered to participate the study. If they accept it as well as their parents, they will be included in the study.

Treatment application will follow recommendations and be realized in out patient clinic with trained nurses.

Tolerance will be assessed by phone call every 24 Hours by investigational team until normalization. Expected duration is less than 24 Hours for 75% patients and 100 % at 72 Hours, from unpublished personal data.

Efficacy will be monitored with usual pain and neuropathic pain tools, adapted to age and cognitive capacities, one month after application.

Treatment may be done three times if needed with a three month interval between each capsaicin patch application.

ELIGIBILITY:
Inclusion Criteria:

* chronic localized neuropathic pain
* capsaicin 8% patch treatment indication validated in a pediatric chronic pain center
* agreement for participation by child and parents

Exclusion Criteria:

* already treated with capsaicin 8% patch in the same body area
* already treated in the same study in an other investigation center
* non willing to participate or parents not willing participation to the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients aged less than 18-y with chronic localized neuropathic pain and capsaicin 8% patch indication validated in a pediatric chronic pain center.
  patient with intellectual development disabilities are accepted
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-09-12 (Estimated)

PRIMARY OUTCOMES:
Success or failure of pain treatment : Number of patients with success and number of patients with failure of treatment with capsaicin | 3 months after last patch application
  The success is defined by the absence of use of pain medication during the three months after the end of capsaicin application protocol

SECONDARY OUTCOMES:
Indication of capsaicin use | At recruitment visit
  Indication for treatment with capsaicine will be collected (context of emergence of pain, descriptive data)
Success or failure of pain treatment : Number of patients who use or not use antalgic and/or comfort medication (including for improving sleep) | Baseline and 1 month, 3 months and 6 months after patch application.
  Use of antalgic and/or comfort medication (including for improving sleep). Success is de fined by the non use of antalgic and/or comfort medication (including for improving sleep)
Neuropathic pain evaluation for child aged from 0 to 4 years | Baseline, 3 months, 6 months and 1 month, 3 months and 6 months after patch application.
  Score of HECP (Hetero-Evaluation of Child Pain) questionnaire, score from 0 to 10 (a higher score means a worse outcome)
Neuropathic pain evaluation for child with intellectual deficiency | Baseline, 3 months, 6 months and 1 month, 3 months and 6 months after patch application.
  Score of PAGID (Pain Assessment Grid - Intellectual Deficiency) or PPP (Pediatric Pain Profile) questionnaire, higher scores are worse outcome
Neuropathic pain description for child aged from 5 to 11 years | Baseline and 1 month, 3 months and 6 months after patch application.
  Global score and subscores of NPSI (Neuropathic Pain Syndrome Inventory), questionnaire with support, score from 0 to 100, higher score is worse outcome
Neuropathic pain diagnostic for child aged from 5 to 11 years | Baseline and 1 month, 3 months and 6 months after patch application.
  Global score of pPN4 (Paediatric Neuropathic Pain 4 points) questionnaire, score from 0 to 10, higher score is worse item
Neuropathic pain evaluation for child aged from 5 to 11 years | Baseline, 3 months, 6 months and 1 month, 3 months and 6 months after patch application.
  Score of pVAS (Paediatric Visual Analogic Scale) or NS (Numeric Scale) or Revised Faces Pain Scales, score from 0 to 10, higher score is worse outcome
Neuropathic pain description for child aged from 12 to 17 years | Baseline and 1 month, 3 months and 6 months after patch application.
  Global score and subscores of NPSI (Neuropathic Pain Syndrome Inventory) questionnaire without support, score from 0 to 100, higher score is worse outcome
Neuropathic pain evaluation for child aged from 12 to 17 years | Baseline, 3 months, 6 months and 1 month, 3 months and 6 months after patch application.
  Score of VAS (Visual Analogic Scale) or NS (Numeric Scale), score from 0 to 10, higher score is worse outcome
Neuropathic pain diagnostic for child aged from 12 to 17 years | Baseline and 1 month, 3 months and 6 months after patch application.
  Global score of NP4 questionnaire (Neuropathic Pain 4 points), score from 0 to 10, higher score is worse item
Functional disability evaluation for child aged from 5 to 17 years | Baseline and 1 month, 3 months and 6 months after patch application.
  Global score of FDI (Functional Disability Inventory) questionnaire, score from 0 to 60, higher score is worse outcome
Pain description for child aged from 5 to 17 years : number of painful access | Baseline and 1 month, 3 months and 6 months after patch application.
  Number of painful access (crisis) in one day
Pain description for child aged from 5 to 17 years : duration of painful access | Baseline and 1 month, 3 months and 6 months after patch application.
  Mean duration of painful access (crisis) in minutes
Pain description for child aged from 5 to 17 years : trigger factor of the painful access | Baseline and 1 month, 3 months and 6 months after patch application.
  Type of trigger factor that leads to the painful access
Pain description for child aged from 5 to 17 years : sensation | Baseline and 1 month, 3 months and 6 months after patch application.
  Description of sensation reported by the child (sensation spontaneously described, qualitative data)
Pain description (observed signs) for child aged from 0 to 4 years or with intellectual deficiency | Baseline and 1 month, 3 months and 6 months after patch application.
  Description of observed signs related to pain
Pain description (sleep quality) for child aged from 0 to 4 years or with intellectual deficiency | Baseline and 1 month, 3 months and 6 months after patch application.
  Description of sleep quality (night awakening / week)
Pain description (child behaviour) for child aged from 0 to 4 years or with intellectual deficiency | Baseline and 1 month, 3 months and 6 months after patch application.
  Description of child behaviour related to pain (antalgic position)
Tolerance assessment (duration of patch application) | Baseline, 3 months and 6 months
  Duration of patch application in minutes
Tolerance assessment (number of patch used) | Baseline, 3 months and 6 months
  Number of patch used during the application
Tolerance assessment (cutaneous state) | Baseline, 3 months and 6 months
  Cutaneous state (burning, erythema, healthy skin, other) just after patch removal
Tolerance assessment (skin aspect) | Baseline, 3 months and 6 months : 4, 8, 24, 48 and 72 hours after patch application
  Local aspect of skin : presence of erythema Yes or No, in the hours and days following patch application
Tolerance assessment (icing) | Baseline, 3 months and 6 months : 4, 8, 24, 48 and 72 hours after patch application
  Need for icing (YES/NO) against pain
Tolerance assessment (rescue medication) | Baseline, 3 months and 6 months : 4, 8, 24, 48 and 72 hours after patch application
  Intake of rescue medication against pain (YES/NO)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe J Le Moine, MD, Principal Investigator — CHRU of Brest
Locations (20):
- France (20):
  - CHU Angers, Angers, France
  - CHU Bordeaux, Bordeaux, France
  - CHR Bourg en Bresse, Bourg-en-Bresse, France
  - CHU de Brest, Brest, France
  - CHU Caen, Caen, France
  - CHU Grenoble, Grenoble, France
  - CHU Lille, Lille, France
  - CHU Limoges, Limoges, France
  - CHU Marseille, Marseille, France
  - CHU Montpellier, Montpellier, France
  - CHU Nancy, Nancy, France
  - CHU Nantes, Nantes, France
  - CHU Robert Debré, Paris, France
  - CHU Trousseau, Paris, France
  - CHU Rouen, Rouen, France
  - CHRU Strasbourg, Strasbourg, France
  - CHU Toulouse, Toulouse, France
  - Institut Gustave Roussy, Villejuif, France
  - CHU d'Amiens, Amiens
  - CHU Lyon, Lyon

IPD SHARING:
Plan to Share IPD: Undecided